CLINICAL TRIAL: NCT04672551
Title: EMDR Treatment in PTSD Following Cardiac Events
Acronym: EMDR_PTSD_MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: EMDR Europe (Industry); Stiftung zur Förderung von Psychiatrie und Psychotherapie (Unknown); EMDR Foundation (Unknown); EMDO Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-00817
Record Dates: First submitted 2020-04-19; First posted 2020-12-17 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Posttraumatic Stress Disorder; Myocardial Infarction; Eye Movement Desensitization and Reprocessing
Keywords: PTSD; MI; ACS; EMDR
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. The efficacy of the standardized trauma-focused procedure in terms of a reduced PTSD symptom level will be tested against a passive waitlist control group.
Who Masked: Outcomes Assessor
Masking Description: Assessors who ascertain the primary outcome variable, i.e. CAPS scores, will be blind to the subject's treatment condition. Randomization will be conducted by a person outside of the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control group (No Intervention): The intervention group consists of 30 patients diagnosed with PTSD induced by ACS. No intervention or any other procedure will be conducted during the study period of 36 weeks. Afterwards these subjects will be offered an EMDR therapy as provided in the intervention.
- Intervention group (Experimental): The intervention group consists of 30 patients diagnosed with PTSD induced by ACS. Eight individual EMDR sessions lasting for 1 hours will be provided over 8 weeks by licensed EMDR therapists from the German-speaking part of Switzerland. Each EMDR session follows a standardized 8-phase protocol.
  Interventions: Behavioral: EMDR Treatment

INTERVENTIONS:
Behavioral: EMDR Treatment — Eight individual EMDR sessions lasting for 1 hours will be provided over 8 weeks by licensed EMDR therapists from the German-speaking part of Switzerland. Each EMDR session follows a standardized 8-phase protocol.
  Arms: Intervention group

SUMMARY:
Cardiac events can often result in debilitating and persistent psychological symptoms. A key question involves whether optimal treatment of cardiac-induced posttraumatic stress disorder (PTSD) reduces PTSD symptoms and thereby may offset the risk of recurrent or worsening cardiovascular disease. Cardiac-induced PTSD 1) is prevalent, 2) features symptoms unique to internal ongoing somatic threat, with fears and worries that can be distinguished from PTSD resulting from external causes, 3) is persistent, 4) is associated with negative physical and emotional consequences, and 5) has not been the subject of randomized-controlled treatment trials (RCT). There is preliminary evidence suggesting that patients with cardiac-disease induced PTSD might particularly profit from EMDR. Nevertheless, this possibility has not been tested in cardiac-induced PTSD. Currently, patients with cardiac-induced PTSD are not routinely offered trauma-focused therapies, with a lack of scientific evidence likely being one major reason for this omission. If our proposed RCT shows that EMDR can be an effective treatment for patients with ACS-induced PTSD, EMDR could be routinely implemented as first-line treatment. The RCT outcomes might inform larger trials to test whether poor prognosis in terms of major adverse cardiovascular events can be improved through EMDR in patients with cardiac-induced PTSD.

DETAILED DESCRIPTION:
There is a lack of research on the efficacy of psychotherapy and especially EMDR in clinical-induced PTSD. In the light of clinical-induced PTSD having different symptoms than traditional PTSD, this lack of research is highly problematic. Specifically, the unique symptom profile in clinical-induced PTSD related to the enduring somatic threat model was not addressed in any of the studies targeting PTSD in cardiac patients. In this regard, EMDR might be most promising: The EMDR protocol includes the assessment of body sensations associated with the target event, which is followed by reprocessing. The bilateral eye movements during reprocessing seem to have de-arousing effects and may thereby interrupt the positive feedback loop between cardiovascular sensations and anxiety-induced arousal as explained by the enduring somatic threat model. Hence, EMDR might be more suitable in cardiac PTSD patients compared to treatment protocols that motivates patients to keep focusing on the traumatic event such as Prolonged Exposure, where higher emotional involvement seems to be related to a better outcome.

Therefore, the here proposed study aims at testing EMDR therapy in c,jj

-induced PTSD in a randomized controlled trial.The here proposed study aims at testing EMDR therapy in ACS-induced PTSD in a randomized controlled trial. More specifically, the efficacy of the standardized trauma-focused procedure in terms of a reduced PTSD symptom level will be tested against a passive waitlist control group.

Intervention group:

The intervention group consists of 30 patients diagnosed with PTSD induced by cardiac events. Eight individual EMDR sessions lasting for 1 hours will be provided over 8 weeks by licensed EMDR therapists from the German-speaking part of Switzerland. Each EMDR session follows a standardized 8-phase protocol. As Shapiro posits that it is necessary to adapt the standard procedures to the unique needs and characteristics of the patient and to apply different EMDR protocols for different pathologies, the therapy for cardiac events was adapted from the standard protocol.

Waiting control group:

The intervention group consists of 30 patients diagnosed with PTSD induced by cardiac events. No intervention or any other procedure will be conducted during the study period of 36 weeks. Afterwards these subjects will be offered an EMDR therapy as provided in the intervention.

Screening for inclusion and exclusion criteria prior to study inclusion:

After discharge, survivors of a cardiac event will be informed about the study by a letter. The Screening will be conducted by phone and/or e-mail. Eligible participants will be screened for inclusion and exclusion criteria. Screening for a probable PTSD diagnosis will be conducted using Part III of the PCL-5 for DSM-5. Subjects who meet a total sum score of 28 or more, will be invited for Baseline a.

Baseline a: Definitive inclusion, baseline measurements, randomization Assessment 1 consists of two appointments taking place at the University Hospital Zurich. During the first appointment, the CAPS-5 and the M.I.N.I will be administered in order to ascertain a PTSD and other psychiatric diagnoses. By means of the CAPS-5, it will be determined whether the participants have PTSD (inclusion criterion and baseline assessment of primary outcome).

As the assessment of the traumatic event during the interview can cause distress (although only minimal and transient), which affects biomarkers, the assessment of cardiovascular biomarkers and stress sensitization by means of the loud-tone procedure will be carried out at a separate appointment.

The second appointment (Baseline b) will be scheduled within 7 days after the first appointment to assess the baseline of all secondary endpoints: 1) saliva and blood samples will be collected to obtain, stress hormones, and cardiovascular biomarkers, including blood pressure; 2) the loud-tone procedure will be administered; 3) patient's medication will be documented. Moreover, the following information will be obtained from the potential participants or from hospital charts: Demographic factors, established cardiovascular risk factors and life style behavior, objective indices of myocardial damage and severity, variables related to patient referral to the coronary care unit, recurrent cardiac symptoms, recurrent hospitalizations, cardiac rehabilitation, doctor visits, pharmacological treatment, adherence to medication, medical comorbidities.

Psychometric data will be collected by means of questionnaires. These questionnaires will be completed during the second appointment or from home via eCRF (Red Cap).

Randomization:

Participants will be randomized into either the intervention group (EMDR treatment) or the wait-list control group. Assessors who ascertain the primary outcome variable, i.e. CAPS scores, will be blind to the subject's treatment condition. Randomization will be conducted by a person outside of the study team.

Intervention period:

After randomization, the intervention (EMDR therapy) will be carried.

Post Treatment and 6-months Follow-up (a/b):

After the intervention (week 12), procedures of assessment 2 related to primary and secondary endpoints (i.e., CAPS, psychophysiological reactivity, psychometry, blood and saliva sampling) will be repeated. In order to test whether the effects of EMDR-treatment are long-lasting, measurements will be repeated at 6-months follow-up. Assessors who ascertain the primary outcome variable, i.e. CAPS scores, will be blind to the subject's treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Men or women
* STEMI (irrespective of troponin, but ST-elevation) or non-STEMI (troponin positive) at the time of the cardiac event, as verified by the cardiologist
* Diagnosis of PTSD caused by the cardiac event

Exclusion Criteria:

* Psychotic disorder, bipolar disorder, substance abuse as measured with the Mini International Neuropsychiatric Interview (M.I.N.I)
* Acute suicidal ideation as assessed with the M.I.N.I.
* Non-selective beta blockers (e.g., propranolol) during the study period
* Ongoing psychological/psychiatric treatment outside of the trial during the study period
* Visionary problems, e.g. strabismus, which does not allow adequate eye movements
* Insufficient knowledge of the German language
* Expected inability or willingness to follow the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Interview-rated posttraumatic stress 3 months Follow-up | 3 months
  The primary endpoint is the interviewer-rated posttraumatic stress level at three months follow-up (by means of the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), with a range from 0-160, whereby higher scores mean a worse outcome).
Interview-rated posttraumatic stress 6 months Follow-up | 6 months
  The primary endpoint is the interviewer-rated posttraumatic stress level at six months follow-up (by means of the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), with a range from 0-160, whereby higher scores mean a worse outcome).

SECONDARY OUTCOMES:
Nose-related psychophysiological stress responses - Heart Rate 3 months | 3 months
  Heart rate (HR)
Nose-related psychophysiological stress responses - Skin Conductance 3 months | 3 months
  skin conductance (SC) responses
Nose-related psychophysiological stress responses - Heart Rate Variability 3 months | 3 months
  Heart rate variability (HRV)
Nose-related psychophysiological stress responses - Heart Rate 6 months | 6 months
  Heart rate (HR)
Nose-related psychophysiological stress responses Skin Conductance - 6 months | 6 months
  skin conductance (SC) responses
Nose-related psychophysiological stress responses - Heart Rate Variability - 6 months | 6 months
  Heart rate variability (HRV)
Stress hormones - Plasma Norepinephrine 3 months | 3 months
  Concentration of Plasma norepinephrine
Stress hormones - Epinephrine 3 months | 3 months
  Concentration of Epinephrine
Stress hormones - Cortisol 3 months | 3 months
  Concentration of Salivary Cortisol
Stress hormones - Plasma Norepinephrine - 6 months | 6 months
  Concentration of Plasma norepinephrine
Stress hormones - Epinephrine 6 months | 6 months
  Concentration of Epinephrine
Stress hormones - Salivary Cortisol 6 months | 6 months
  Concentration of Salivary Cortisol
Cardiometabolic biomarkers - metabolic factors 3 months | 3 months
  Metabolic Factors (Concentration of total cholesterol, low density lipoprotein (LDL-C), high density lipoprotein (HDL-C), triglycerides and glucose)
Cardiometabolic biomarkers - metabolic factors 6 months | 6 months
  Metabolic Factors (Concentration of total cholesterol, low density lipoprotein (LDL-C), high density lipoprotein (HDL-C), triglycerides and glucose)
Cardiometabolic biomarkers - inflammation markers 3 months | 3 months
  Inflammation markers (Concentration of high-sensitive C-reactive protein (hs-CRP), Interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha))
Cardiometabolic biomarkers - inflammation markers 6 months | 6 months
  Inflammation markers (Concentration of high-sensitive C-reactive protein (hs-CRP), Interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha))

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mueller-Pfeiffer, PD Dr. med., Principal Investigator — University of Zurich/University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT04672551/Prot_SAP_000.pdf